CLINICAL TRIAL: NCT01397552
Title: A Prospective, Randomized, Double-Blind Study to Compare the Effects of Dexamethasone Versus Depo-Medrol When Used in Lumbar Epidural Injections
Brief Title: Dexamethasone Versus Depo Medrol in Lumbar Epidurals
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment, too many subjects getting second injection
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, William Lavelle, Associate Professor, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB 5824
Record Dates: First submitted 2011-07-15; First posted 2011-07-19 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2018-10

CONDITIONS: Lumbar Spine Disc Herniation; Lumbar Radiculitis; Lumbar Back Pain
MeSH Terms: conditions — Radiculopathy; Low Back Pain | interventions — Dexamethasone; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Active Comparator): Subjects randomized to receive dexamethasone, will undergo epidural using this medication, however the physician and subject will be blinded
  Interventions: Drug: Dexamethasone
- methylprednisolone acetate (Active Comparator): Subjects randomized to receive methylprednisolone acetate, will undergo epidural using this medication, however the physician and subject will be blinded
  Interventions: Drug: methylprednisolone acetate

INTERVENTIONS:
Drug: Dexamethasone — 10 mg/mL injected into lumbar spine, one level, one injection
  Other Names: dexpak
  Arms: Dexamethasone
Drug: methylprednisolone acetate — 80 mg of methylprednisolone acetate will be given in the lumbar spine, one level, one time
  Other Names: Depo-Medrol
  Arms: methylprednisolone acetate

SUMMARY:
Comparison of Dexamethasone versus Depo Medrol when used in lumbar epidural injections will be conducted on subjects that have not had previous injections or have not had an injection in the last 12 months. Subjects must be receiving one level injection and not had prior surgery at that level.

DETAILED DESCRIPTION:
Central Epidural Steroid Injections (ESI) and Selective Nerve Root Blocks (SNRB) are often used for the non-surgical treatment of lumbar disc herniations and lumbar radiculitis (radiating pain). Numerous authors have reported on their value in treating patients with radicular pain with the possibility of delaying or even obviating the need for surgery in well-selected patients.. There are two well-performed clinical studies in the peer-reviewed medical literature that specifically examined the crossover rates to surgery for patients who received either ESI or SNRB. In a prospective study, Buttermann et al. found a crossover rate to surgery for patients with symptomatic disc herniations treated with ESI of 54% (27/50) . In a separate prospective study, Riew et al. followed patients after selective nerve root blocks and found that similarly 53% (29/55) of their patients had avoided surgery after a selective nerve root block during their initial follow-up of 13-28 months. In a later study that followed that same population, 76% (16/21) of those patients who had avoided surgery at one year still avoided surgery at a minimum of five year follow-up.

Epidural steroid injections are a common treatment option for patients with disc herniations and radiating leg pain. They have been used for low back problems since 1922 and are still an integral part of the non-surgical management of a variety of spine related problems. The goal of the injection is reduction in pain, increased quality of life and increased function.

Most practitioners will agree that, while the effects of the injection tend to be temporary-providing relief from pain for one week up to one year-an epidural can be very beneficial for a patient during an acute episode of back and/or leg pain. Importantly, an injection can provide sufficient pain relief to allow a patient to progress with a rehabilitative stretching and exercise program.

Many previous studies on epidural injections did not include use of fluoroscopy or xray to verify proper placement of the medication despite the fact that fluoroscopic guidance is routinely used today. Additionally, many studies do not classify patients according to diagnosis and tend to "lump" different types, sources of pain together.

Commonly used steroid preparations include betamethasone, triamcinolone, dexamethasone and methylprednisolone. Unfortunately, there is no consensus regarding the most effective medication, dose, volume or frequency used for ESIs.

This investigator-initiated study is being conducted to compare the effects of epidural injections on low back pain when using either dexamethasone or methylprednisolone (Depo-Medrol). The physicians listed would like to compare these two medications to assess if one is more effective than the other. Both medications are FDA approved and are not experimental.

Dexamethasone is the only nonparticulate corticosteroid, has a rapid onset that acts as an anti-inflammatory and immunosuppressant.

Depo-Medrol is a synthetic steroid (cortisone) medication which also acts as an anti-inflammatory when physicians administer an epidural for relief of low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic low back pain of radicular origin of > 4 weeks but < 6 months
2. Failure of conservative therapy to include physical therapy and pharmacotherapy
3. Patient is at least 21 years of age
4. Patient is willing to be blinded to treatment until after the 12 week post injection visit.
5. Patient is willing and able to review and sign the study informed consent form.

Exclusion Criteria:

1. Patient has a mental or physical condition that would invalidate evaluation results.
2. Patient has had prior lumbar surgery at any level.
3. Patient is scheduled to have more than one level of steroid injection.
4. Patient is pregnant
5. Patient has systemic infection at the proposed injection site
6. Patient has osteopenia osteoporosis, or osteomalacia
7. Patient has a disease of bone metabolism
8. Patient has history of renal insufficiency or kidney disease of any kind
9. Patient is undergoing chemotherapy or radiation treatment
10. Patient is currently involved in a study of another product for similar purpose
11. Patient requires post op management with NSAIDS
12. Patient has know allergy to corticosteroids, contrast dye or anesthetics
13. Patient is unable to speak/read English
14. Patient is a prisoner

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suehun Ho, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- Upstate Orthpedics, East Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone | Methylprednisolone Acetate
Started | 4 | 4
Completed | 1 | 3
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: analysis was not sstarted as enrollment was too low and half of the subjects did not complete the study requirements, no data was collected for analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Methylprednisolone Acetate | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous [unit: years]
Sex: Female, Male
Region of Enrollment

OUTCOME MEASURES:

1. Primary Outcome: To Determine if One Medication is Better at Relieving Pain Than the Other.
Description: Subjects will be asked to return at 2 wks, 6 wks and 12 weeks the above time points to complete outcome measurements questionnaires and undergo a neurological examination, the 12 weeks outcome should show improvement s/p injection
Time Frame: 12 wk post injection
Population: enrollment was too low and half of the subjects did not complete study requirements, no data collected for analysis
Arm/Group | Dexamethasone | Methylprednisolone Acetate
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dexamethasone | Methylprednisolone Acetate
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No